CLINICAL TRIAL: NCT03641586
Title: A Phase I, Single and Multiple Dose Escalation/Expansion Study to Investigate the Safety, Tolerability, Pharmacokinetics, Food Effect, and Preliminary Antitumor Activities of BGB-283 in Chinese Subjects With Local Advanced or Metastatic Malignant Solid Tumor
Brief Title: The Study of BGB-283 in Chinese Subjects With Local Advanced or Metastatic Malignant Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-283-CN-001; CTR20150575 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2018-07-11; First posted 2018-08-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors
Keywords: Dose Escalation; Dose Expansion; BGB-283
MeSH Terms: interventions — BGB-283

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stage I (Experimental): Approximately 25-35 Chinese subjects with local advanced or metastatic malignant solid tumor will be enrolled in the dose escalation stage of BGB-283 until maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) determination
  Interventions: Drug: BGB-283
- Stage II (Experimental): Approximately 15-30 melanoma subjects will be enrolled in dose expansion stage of BGB-283
  Interventions: Drug: BGB-283
- Stage III (Experimental): 20 subjects will be enrolled for food effect stage of BGB-283
  Interventions: Drug: BGB-283

INTERVENTIONS:
Drug: BGB-283

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, food effect, and preliminary antitumor activities of BGB-283 in Chinese subjects with local advanced or metastatic malignant solid tumor.

DETAILED DESCRIPTION:
"This study is conducted on the basis of the completed multi-dose, dose escalation, Phase IA trial in Australia, is a dose-finding, dose expansion and food effects study of BGB-283 capsules in Chinese patients with locally advanced or metastatic solid tumor to determine the tolerability, safety, pharmacokinetic profiles, preliminary efficacy, food effects under high-fat meal on the absorption and metabolism of BGB-283, and preliminary anti-tumor efficacy.

The study was conducted in three phases: Stage I for dose escalation, Stage II for dose expansion and Stage III for food effects on pharmacokinetics under high fat meal.

Stage I Dose escalation: In a open-label, dose-escalation design, dose escalation will be performed with the '3 + 3' scheme and the dosage levels of BGB-283 capsules will be gradually increased.

Stage II Dose expansion: 20 mg/qd and 30 mg/qd are considered as effective and safe doses, based on preliminary results from Phase IA clinical studies in Australia. To further understand the preliminary pharmacodynamic results of BGB-283 in Chinese patients with malignant melanoma, 20mg/qd dose expansion study in B-RAF mutated malignant melanoma will be further explored if it has been proved to be a safe dose in Chinese population according to the '3 + 3' scheme.

Stage III uses multi-center, open, two-group crossover self-control design to compare the high-fat meal effect on pharmacokinetics."

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent prior to enrollment.
2. Male or female and between 18 and 75 years old.
3. A life expectancy of more than 12 weeks.
4. Stage I and III: Histologically or cytologically confirmed advanced or metastatic solid tumor for which no effective standard therapy is available. We simultaneously require patients with one of B-RAF, N-RAS, or K-RAS mutation positive solid tumor.
5. In Stage II: we require advanced or metastatic melanoma with the B-RAF mutation.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
7. Able to swallow and retain oral medication.
8. Adequate bone marrow, liver, and renal function:

   * Hemoglobin > 90 g/L
   * Absolute neutrophil count ≥ 1.5x10^9/L
   * Platelets ≥ 100 x10^9/L
   * Total bilirubin ≤1.5 times the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with known liver metastasis)
   * Creatinine clearance ≥ 50 mL/min (calculated by the Cockcroft Gault formula).

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. Prior chemotherapy, radiotherapy, immunotherapy or any investigational therapies used to control cancer must have been completed at least 4 weeks or at least 5 half-lives (whichever is shorter before study drug administration, but at least 21 days)
3. Any major surgery within 28 days prior to enrollment.
4. Any radiotherapy for metastatic foci within 14 days prior to enrollment,
5. Unresolved toxicity > Grade 1 (according to NCI-CTCAE, Version 4.03) from previous anti cancer therapy.
6. History or presence of gastrointestinal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
7. Any clinical significant active infection that need systematic treatment, including HIV positive subjects, or known Hepatitis B or C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Stage 1: Number of participants with treatment-related adverse events as assessed by CTC AE 4.03, 1 year in average | From signing the informed consent form and throughout the study, 1 year in average
Stage 2: To determine the objective response rate (ORR) as assessed by RECIST, Version 1.1 | Every 6 weeks from first dose until the date of first documented progression or date of death from any cause, whichever came first, 1 year in average
Stage 3: Area under the plasma concentration-time curve from time 0 to infinity time (AUC) | Within 43 days since first dose
Stage 3: Maximum plasma concentration (Cmax) | Within 43 days since first dose
Stage 3: Terminal elimination half-life (t1/2) | Within 43 days since first dose
Stage 3: Detect Ka for Pop-PK analysis | Within 43 days since first dose
Stage 3: Detect CL/F for Pop-PK analysis | Within 43 days since first dose
Stage 3: Detect Vc/F for Pop-PK analysis | Within 43 days since first dose

SECONDARY OUTCOMES:
Stage 1: Area under the plasma concentration-time curve from time 0 to infinity time (AUC) | Within 43 days since first dose
Stage 1: Maximum plasma concentration (Cmax) | Within 43 days since first dose
Stage 1: Terminal elimination half-life (t1/2) | Within 43 days since first dose
Stage 1: To determine the objective response rate (ORR) as assessed by RECIST, Version 1.1 | Every 6 weeks from first dose until the date of first documented progression or date of death from any cause, whichever came first, 1 year in average
Stage 2: Number of participants with treatment-related adverse events as assessed by CTC AE 4.03, 1 year in average | From signing the informed consent form and throughout the study, 1 year in average
Stage 3: To determine the objective response rate (ORR) as assessed by RECIST, Version 1.1 | Every 6 weeks from first dose until the date of first documented progression or date of death from any cause, whichever came first, 1 year in average

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Li, MD, Study Director — BeiGene
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China